CLINICAL TRIAL: NCT07081243
Title: A Prospective, Single-group, Non-interventional, Non-blinded, Observational Study to Evaluate the Long-term Safety, Efficacy, and Durability of Symplicity Spyral Renal Denervation System in China
Brief Title: Symplicity China Study
Status: Recruiting | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT24050
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Symplicity Spyral Renal Denervation System — Symplicity Renal Denervation

SUMMARY:
The Symplicity China study will evaluate the real-world long-term safety, efficacy, and durability of the Symplicity Spyral system in a population of approximately 500 renal denervation treated subjects with up to 36 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Patients diagnosed with resistant hypertension or antihypertensive drug intolerance and treated with Symplicity Spyral Renal Denervation System. Resistant hypertension, defined as having an office systolic blood pressure (SBP) ≥140 mmHg despite appropriate lifestyle measures and being treated with three or more antihypertensive medications (including a diuretic) for more than 3 months; or drug intolerance, defined as patients who cannot tolerate medication due to contraindications or adverse effects.
3. The patient voluntarily undergoes renal denervation; the patient has been informed of the observational nature of the study; the patient voluntarily provides written informed consent ("Patient Informed Consent Form") and willingly participates in the study.

Exclusion Criteria:

1. At least one main renal artery with a diameter less than 3 mm or greater than 8 mm.
2. Presence of fibromuscular dysplasia.
3. Renal artery stent placement within 3 months prior to the procedure.
4. Presence of Renal artery aneurysms.
5. Presence of more than 50% stenosis in any treatable vessel.
6. Pregnant.
7. Present of renal or adrenal tumors.
8. Iliac/femoral artery stenosis prevents catheter insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with resistant hypertension or antihypertensive drug intolerance.
  Resistant hypertension, defined as having an office systolic blood pressure (SBP) ≥140 mmHg despite appropriate lifestyle measures and being treated with three or more antihypertensive medications (including a diuretic) for more than 3 months.
  Drug intolerance, defined as patients who cannot tolerate medication due to contraindications or adverse effects.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: Change in systolic blood pressure (SBP) from baseline to 6 months post-procedure as measured by office blood pressure. | 6 months post-procedure

SECONDARY OUTCOMES:
Changes in office blood pressure | 1, 3, 6, 12, 24 and 36 months post-procedure
Changes in home blood pressure | 1, 3, 6, 12, 24 and 36 months post-procedure
Changes in 24-hour ambulatory blood pressure | 1, 3, 6, 12, 24 and 36 months post-procedure
Changes of Number of medications | 1, 3, 6, 12, 24 and 36 months post-procedure
Changes of Medication burden | 1, 3, 6, 12, 24 and 36 months post-procedure
Proportion of subjects achieving blood pressure reduction and control to ≤140 mmHg (measured by OBP, HBP, and ABPM) | 1, 3, 6, 12, 24 and 36 months post-procedure
Event rates | 1, 3, 6, 12, 24 and 36 months post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China